CLINICAL TRIAL: NCT01365520
Title: Multi-Centre, Open-Label, Randomised Trial Investigating the Pharmacokinetics of a Single Dose of NNC 0155-0000-0004 (N8) in Patients With Haemophilia A
Brief Title: A Single Dose Trial of NNC 0155-0000-0004 in Patients With Haemophilia A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-3893; 2010-023921-39 (EudraCT Number); U1111-1118-2228 (Other: WHO)
Record Dates: First submitted 2011-05-30; First posted 2011-06-03 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N8 (Experimental)
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — A single dose will be administered i.v. (into the vein). Subjects will be randomised to one of two lots of NNC 0155-0000-0004.

SUMMARY:
This trial is conducted in Asia and Europe. The aim of the trial is to investigate the pharmacokinetics (the rate at which the trial drug is eliminated from the body) of a single dose of turoctocog alfa (NNC 0155-0000-0004 (N8)) in patients with haemophilia A. Participation in this trial is dependent on previous participation in trial NN7008-3543 (Part B) (NCT00840086).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the diagnosis of severe haemophilia A (factor VIII less than or equal to 1%)
* Body weight between 10 to 120 kg
* Subjects who have completed NN7008-3543 (Part B) or subjects participating in NN7008-3568 after completion of NN7008-3543 (NCT00840086)

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Previous participation in this trial defined as withdrawal
* Planned surgery during the trial period (catheter, stents, ports, and dental extractions do not count as surgeries and will not exclude the subject)
* Any disease or condition which, according to the trial physician's judgement, could imply a potential hazard to the subject, interfere with the trial participation or trial outcome

Ages: 12 Years to 56 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve | Infusion, 48 hours
Incremental recovery | Infusion, 30 minutes
In vivo t1/2 | Infusion, 48 hours
Total clearance (CL) | Infusion, 48 hours

SECONDARY OUTCOMES:
Maximal concentration (Cmax) | 15 minutes after trial drug administration
Number of adverse events | up to 48 hours after trial drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, London, United Kingdom

REFERENCES:
- [Result] Jimenez-Yuste V, Lejniece S, Klamroth R, Suzuki T, Santagostino E, Karim FA, Saugstrup T, Moss J. The pharmacokinetics of a B-domain truncated recombinant factor VIII, turoctocog alfa (NovoEight(R)), in patients with hemophilia A. J Thromb Haemost. 2015 Mar;13(3):370-9. doi: 10.1111/jth.12816. Epub 2015 Feb 13. PMID 25495795
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com